CLINICAL TRIAL: NCT00095238
Title: Irbesartan in Heart Failure With Preserved Systolic Function (I-Preserve)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV131-148
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Results first posted 2010-06-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Irbesartan
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irbesartan — Tablets, Oral, titration from 75 to 300 mg, once daily up to 6 years
  Arms: 1
Drug: Placebo — Tablets, Oral, titration from 75 to 300 mg, once daily up to 6 years
  Arms: 2

SUMMARY:
The purpose of this clinical research study is to learn if Irbesartan is superior to placebo in reducing mortality and cardiovascular morbidity in subjects with heart failure with preserved systolic function. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age >= 60 years with current symptoms of heart failure consistent with New York Heart Association (NYHA) class II-IV
* Left ventricular ejection fraction (LVEF) > = 45%
* Willing to provide written informed consent AND hospitalization for heart failure within the past 6 months OR various abnormalities in electrocardiogram, echocardiogram or chest x-ray indicating heart disease.

Exclusion Criteria:

* Acute myocardial infarction within 3 months;
* Heart revascularization procedure within 3 months;
* Hospitalization for angina within 3 months;
* Other heart surgery
* Life-threatening or uncontrolled arrhythmia
* Subjects with an implantable cardioverter-defibrillator that has discharged in the past 3 months;
* Stroke or surgery of the arteries in the brain within 3 months;
* Serious lung disease which requires use of home oxygen.
* Significantly low blood pressure
* Significantly high blood pressure
* Other known diseases that may limit life expectancy to <3 years;
* Known or suspected bilateral kidney artery narrowing;
* Geographic or social factors making study participation and follow-up impractical.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4128 (Actual)
Dates: Start 2002-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (229):
- United States (60):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Peoria, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Los Angeles, California
  - Local Institution, San Diego, California
  - Local Institution, San Francisco, California
  - Local Institution, Farmington, Connecticut
  - Local Institution, Jacksonville, Florida
  - Local Institution, Jacksonville Beach, Florida
  - Local Institution, Lake Worth, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Vero Beach, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Peoria, Illinois
  - Local Institution, Jeffersonville, Indiana
  - Local Institution, Louisville, Kentucky
  - Local Institution, Chalmette, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Auburn, Maine
  - Local Institution, Takoma Park, Maryland
  - Local Institution, Towson, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Haverhill, Massachusetts
  - Local Institution, Natick, Massachusetts
  - Local Institution, Detroit, Michigan
  - Local Institution, Petoskey, Michigan
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Reno, Nevada
  - Local Institution, Lebanon, New Hampshire
  - Local Institution, Elmer, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Albany, New York
  - Local Institution, East Syracuse, New York
  - Local Institution, Flushing, New York
  - Local Institution, Rochester, New York
  - Local Institution, The Bronx, New York
  - Local Institution, Troy, New York
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Concord, North Carolina
  - Local Institution, Durham, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Canton, Ohio
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Lorain, Ohio
  - Local Institution, Sandusky, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Flourtown, Pennsylvania
  - Local Institution, Lancaster, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Germantown, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Lynchberg, Virginia
  - Local Institution, Richmond, Virginia
  - Local Institution, South Boston, Virginia
  - Local Institution, Spokane, Washington
  - Local Institution, Madison, Wisconsin
- Argentina (6):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, Corrientes, Corrientes Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Mendoza, Mendoza Province
  - Local Institution, Rosario, Santa Fe Province
- Australia (11):
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Concord, New South Wales
  - Local Institution, Garran, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Auchenflower, Queensland
  - Local Institution, Brisbane, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Launceston, Tasmania
  - Local Institution, Geelong, Victoria
  - Local Institution, Prahran, Victoria
- Belgium (9):
  - Local Institution, Aalst
  - Local Institution, Aye
  - Local Institution, Borgerhout
  - Local Institution, Genk-waterschei
  - Local Institution, Ghent
  - Local Institution, Hasselt
  - Local Institution, Huy
  - Local Institution, Leuven
  - Local Institution, Verviers
- Brazil (6):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Goiania-go, Goiás
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, Sao Paulo, Sp, São Paulo
- Canada (12):
  - Local Institution, Calgary, Alberta
  - Local Institution, Victoria, British Columbia
  - Local Institution, Ajax, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, Rexdale, Ontario
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Weston, Ontario
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Ste-Foy, Quebec
- Czechia (2):
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
- Denmark (2):
  - Local Institution, Copenhagen
  - Local Institution, Copenhagen Nv
- France (17):
  - Local Institution, Abbeville
  - Local Institution, Cholet
  - Local Institution, Dax
  - Local Institution, Gap
  - Local Institution, Langres
  - Local Institution, Lille
  - Local Institution, Montbéliard
  - Local Institution, Paris
  - Local Institution, Poissy
  - Local Institution, Pontoise
  - Local Institution, Provins
  - Local Institution, Roubaix
  - Local Institution, Rouen
  - Local Institution, St-Malo
  - Local Institution, Tours
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution, Vichy
- Germany (16):
  - Local Institution, Bad Homburg
  - Local Institution, Berlin
  - Local Institution, Göttingen
  - Local Institution, Gunzenhausen
  - Local Institution, Halle
  - Local Institution, Homburg / Saar
  - Local Institution, Jena
  - Local Institution, Langen
  - Local Institution, Leipzig
  - Local Institution, Mainz
  - Local Institution, Marburg
  - Local Institution, München
  - Local Institution, Regensburg
  - Local Institution, Stuttgart
  - Local Institution, Witten
  - Local Institution, Würzburg
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Pátrai
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Siófok
  - Local Institution, Szeged
- Ireland (2):
  - Local Institution, County Dublin, Dublin
  - Local Institution, Dublin, Dublin
- Italy (11):
  - Local Institution, Ascoli Piceno
  - Local Institution, Bologna
  - Local Institution, Brescia
  - Local Institution, Cosenza
  - Local Institution, Pavia
  - Local Institution, Perugia
  - Local Institution, Piacenza
  - Local Institution, Roma
  - Local Institution, Siena
  - Local Institution, Trieste
  - Local Institution, Udine
- Mexico (4):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, San Pedro Garza García, Nuevo León
- Netherlands (20):
  - Local Institution, Alkmaar
  - Local Institution, Almere Stad
  - Local Institution, Amersfoort
  - Local Institution, Apeldoorn
  - Local Institution, Assen
  - Local Institution, Breda
  - Local Institution, Delft
  - Local Institution, Emmen
  - Local Institution, Gorinchem
  - Local Institution, Groningen
  - Local Institution, Heemstede
  - Local Institution, Helmond
  - Local Institution, Hengelo Ov
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
  - Local Institution, Sittard
  - Local Institution, Sneek
  - Local Institution, Veldhoven
  - Local Institution, Vlaardingen
  - Local Institution, Zaandam
- Norway (3):
  - Local Institution, Baerum Postterminal
  - Local Institution, Stavanger
  - Local Institution, Tønsberg
- Poland (6):
  - Local Institution, Bydgoszcz
  - Local Institution, Katowice
  - Local Institution, Piotrkow Tryb.
  - Local Institution, Stalowa Wola
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Portugal (2):
  - Local Institution, Lisbon
  - Local Institution, Matosinhos Municipality
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
- South Africa (5):
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Morningside, Gauteng
  - Local Institution, Parktown West, Gauteng
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, KwaKhangela, KwaZulu-Natal
- Spain (10):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Córdoba
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Murcia
  - Local Institution, Palma de Mallorca
  - Local Institution, Seville
  - Local Institution, Valencia
  - Local Institution, Zaragoza
- Sweden (7):
  - Local Institution, Falun
  - Local Institution, Gothenburg
  - Local Institution, Linköping
  - Local Institution, Malmo
  - Local Institution, Skellefteå
  - Local Institution, Stockholm
  - Local Institution, Sundsvall
- Switzerland (3):
  - Local Institution, Bellinzona
  - Local Institution, Liestal
  - Local Institution, Zurich
- United Kingdom (6):
  - Local Institution, Glasgow, Dumbartonshire
  - Local Institution, Romford, Essex
  - Local Institution, Londonderry, Londonderry
  - Local Institution, Hull, Yorkshire
  - Local Institution, York, Yorkshire
  - Local Institution, Dundee

REFERENCES:
- [Result] Massie BM, Carson PE, McMurray JJ, Komajda M, McKelvie R, Zile MR, Anderson S, Donovan M, Iverson E, Staiger C, Ptaszynska A; I-PRESERVE Investigators. Irbesartan in patients with heart failure and preserved ejection fraction. N Engl J Med. 2008 Dec 4;359(23):2456-67. doi: 10.1056/NEJMoa0805450. Epub 2008 Nov 11. PMID 19001508
- [Result] Zile MR, Gaasch WH, Anand IS, Haass M, Little WC, Miller AB, Lopez-Sendon J, Teerlink JR, White M, McMurray JJ, Komajda M, McKelvie R, Ptaszynska A, Hetzel SJ, Massie BM, Carson PE; I-Preserve Investigators. Mode of death in patients with heart failure and a preserved ejection fraction: results from the Irbesartan in Heart Failure With Preserved Ejection Fraction Study (I-Preserve) trial. Circulation. 2010 Mar 30;121(12):1393-405. doi: 10.1161/CIRCULATIONAHA.109.909614. Epub 2010 Mar 15. PMID 20231531
- [Result] McMurray JJ, Carson PE, Komajda M, McKelvie R, Zile MR, Ptaszynska A, Staiger C, Donovan JM, Massie BM. Heart failure with preserved ejection fraction: clinical characteristics of 4133 patients enrolled in the I-PRESERVE trial. Eur J Heart Fail. 2008 Feb;10(2):149-56. doi: 10.1016/j.ejheart.2007.12.010. PMID 18279770
- [Result] Carson P, Massie BM, McKelvie R, McMurray J, Komajda M, Zile M, Ptaszynska A, Frangin G; I-PRESERVE Investigators. The irbesartan in heart failure with preserved systolic function (I-PRESERVE) trial: rationale and design. J Card Fail. 2005 Oct;11(8):576-85. doi: 10.1016/j.cardfail.2005.06.432. PMID 16230259
- [Result] McKelvie RS, Komajda M, McMurray J, Zile M, Ptaszynska A, Donovan M, Carson P, Massie BM; I-Preserve Investigators. Baseline plasma NT-proBNP and clinical characteristics: results from the irbesartan in heart failure with preserved ejection fraction trial. J Card Fail. 2010 Feb;16(2):128-34. doi: 10.1016/j.cardfail.2009.09.007. Epub 2009 Nov 4. PMID 20142024
- [Derived] Lassen MCH, Ostrominski JW, Claggett BL, Neuen BL, Beldhuis IE, Butt JH, Biering-Sorensen T, Desai AS, Lewis EF, Jhund PS, Mc Causland F, Anand IS, Pfeffer MA, Pitt B, Zannad F, Zile MR, McMurray JJV, Solomon SD, Vaduganathan M. Obesity and Risk of Kidney Outcomes in Heart Failure With Preserved Ejection Fraction: A Participant-Level Pooled Analysis of 4 Contemporary Trials. JACC Heart Fail. 2025 Aug;13(8):102498. doi: 10.1016/j.jchf.2025.03.042. Epub 2025 Jun 9. PMID 40494011
- [Derived] Kondo T, Campbell R, Jhund PS, Anand IS, Carson PE, Lam CSP, Shah SJ, Vaduganathan M, Zannad F, Zile MR, Solomon SD, McMurray JJV. Low Natriuretic Peptide Levels and Outcomes in Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2024 Aug;12(8):1442-1455. doi: 10.1016/j.jchf.2024.04.027. Epub 2024 Jun 19. PMID 38904646
- [Derived] Kondo T, Dewan P, Anand IS, Desai AS, Packer M, Zile MR, Pfeffer MA, Solomon SD, Abraham WT, Shah SJ, Lam CSP, Jhund PS, McMurray JJV. Clinical Characteristics and Outcomes in Patients With Heart Failure: Are There Thresholds and Inflection Points in Left Ventricular Ejection Fraction and Thresholds Justifying a Clinical Classification? Circulation. 2023 Aug 29;148(9):732-749. doi: 10.1161/CIRCULATIONAHA.122.063642. Epub 2023 Jun 27. PMID 37366061
- [Derived] Kondo T, Jering KS, Jhund PS, Anand IS, Desai AS, Lam CSP, Maggioni AP, Martinez FA, Packer M, Petrie MC, Pfeffer MA, Redfield MM, Rouleau JL, van Veldhuisen DJ, Zannad F, Zile MR, Solomon SD, McMurray JJV. Predicting Stroke in Heart Failure and Preserved Ejection Fraction Without Atrial Fibrillation. Circ Heart Fail. 2023 Jul;16(7):e010377. doi: 10.1161/CIRCHEARTFAILURE.122.010377. Epub 2023 Jun 23. PMID 37350280
- [Derived] Curtain JP, Adamson C, Kondo T, Butt JH, Desai AS, Zannad F, Rouleau JL, Rohde LE, Kober L, Anand IS, van Veldhuisen DJ, Zile MR, Lefkowitz MP, Solomon SD, Packer M, Petrie MC, Jhund PS, McMurray JJV. Investigator-reported ventricular arrhythmias and mortality in heart failure with mildly reduced or preserved ejection fraction. Eur Heart J. 2023 Feb 21;44(8):668-677. doi: 10.1093/eurheartj/ehac801. PMID 36632831
- [Derived] Shen L, Jhund PS, Anand IS, Carson PE, Desai AS, Granger CB, Kober L, Komajda M, McKelvie RS, Pfeffer MA, Solomon SD, Swedberg K, Zile MR, McMurray JJV. Developing and validating models to predict sudden death and pump failure death in patients with heart failure and preserved ejection fraction. Clin Res Cardiol. 2021 Aug;110(8):1234-1248. doi: 10.1007/s00392-020-01786-8. Epub 2020 Dec 10. PMID 33301080
- [Derived] Tromp J, Shen L, Jhund PS, Anand IS, Carson PE, Desai AS, Granger CB, Komajda M, McKelvie RS, Pfeffer MA, Solomon SD, Kober L, Swedberg K, Zile MR, Pitt B, Lam CSP, McMurray JJV. Age-Related Characteristics and Outcomes of Patients With Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2019 Aug 6;74(5):601-612. doi: 10.1016/j.jacc.2019.05.052. PMID 31370950
- [Derived] Kristensen SL, Mogensen UM, Jhund PS, Rorth R, Anand IS, Carson PE, Desai AS, Pitt B, Pfeffer MA, Solomon SD, Zile MR, Kober L, McMurray JJV. N-Terminal Pro-B-Type Natriuretic Peptide Levels for Risk Prediction in Patients With Heart Failure and Preserved Ejection Fraction According to Atrial Fibrillation Status. Circ Heart Fail. 2019 Mar;12(3):e005766. doi: 10.1161/CIRCHEARTFAILURE.118.005766. PMID 30871349
- [Derived] Kristensen SL, Mogensen UM, Jhund PS, Petrie MC, Preiss D, Win S, Kober L, McKelvie RS, Zile MR, Anand IS, Komajda M, Gottdiener JS, Carson PE, McMurray JJ. Clinical and Echocardiographic Characteristics and Cardiovascular Outcomes According to Diabetes Status in Patients With Heart Failure and Preserved Ejection Fraction: A Report From the I-Preserve Trial (Irbesartan in Heart Failure With Preserved Ejection Fraction). Circulation. 2017 Feb 21;135(8):724-735. doi: 10.1161/CIRCULATIONAHA.116.024593. Epub 2017 Jan 4. PMID 28052977
- [Derived] Gandhi PU, Chow SL, Rector TS, Krum H, Gaggin HK, McMurray JJ, Zile MR, Komajda M, McKelvie RS, Carson PE, Januzzi JL Jr, Anand IS. Prognostic Value of Insulin-Like Growth Factor-Binding Protein 7 in Patients with Heart Failure and Preserved Ejection Fraction. J Card Fail. 2017 Jan;23(1):20-28. doi: 10.1016/j.cardfail.2016.06.006. Epub 2016 Jun 16. PMID 27317843
- [Derived] Badar AA, Perez-Moreno AC, Hawkins NM, Jhund PS, Brunton AP, Anand IS, McKelvie RS, Komajda M, Zile MR, Carson PE, Gardner RS, Petrie MC, McMurray JJ. Clinical Characteristics and Outcomes of Patients With Coronary Artery Disease and Angina: Analysis of the Irbesartan in Patients With Heart Failure and Preserved Systolic Function Trial. Circ Heart Fail. 2015 Jul;8(4):717-24. doi: 10.1161/CIRCHEARTFAILURE.114.002024. Epub 2015 Jun 11. PMID 26067854
- [Derived] Oluleye OW, Rector TS, Win S, McMurray JJ, Zile MR, Komajda M, McKelvie RS, Massie B, Carson PE, Anand IS. History of atrial fibrillation as a risk factor in patients with heart failure and preserved ejection fraction. Circ Heart Fail. 2014 Nov;7(6):960-6. doi: 10.1161/CIRCHEARTFAILURE.114.001523. Epub 2014 Sep 15. PMID 25225241
- [Derived] Bohm M, Perez AC, Jhund PS, Reil JC, Komajda M, Zile MR, McKelvie RS, Anand IS, Massie BM, Carson PE, McMurray JJ; I-Preserve Committees and Investigators. Relationship between heart rate and mortality and morbidity in the irbesartan patients with heart failure and preserved systolic function trial (I-Preserve). Eur J Heart Fail. 2014 Jul;16(7):778-87. doi: 10.1002/ejhf.85. Epub 2014 May 23. PMID 24864045
- [Derived] Lam CS, Carson PE, Anand IS, Rector TS, Kuskowski M, Komajda M, McKelvie RS, McMurray JJ, Zile MR, Massie BM, Kitzman DW. Sex differences in clinical characteristics and outcomes in elderly patients with heart failure and preserved ejection fraction: the Irbesartan in Heart Failure with Preserved Ejection Fraction (I-PRESERVE) trial. Circ Heart Fail. 2012 Sep 1;5(5):571-8. doi: 10.1161/CIRCHEARTFAILURE.112.970061. Epub 2012 Aug 10. PMID 22887722
- [Derived] Rector TS, Carson PE, Anand IS, McMurray JJ, Zile MR, McKelvie RS, Komajda M, Kuskowski M, Massie BM; I-PRESERVE Trial Investigators. Assessment of long-term effects of irbesartan on heart failure with preserved ejection fraction as measured by the minnesota living with heart failure questionnaire in the irbesartan in heart failure with preserved systolic function (I-PRESERVE) trial. Circ Heart Fail. 2012 Mar 1;5(2):217-25. doi: 10.1161/CIRCHEARTFAILURE.111.964221. Epub 2012 Jan 20. PMID 22267751
- [Derived] Zile MR, Gottdiener JS, Hetzel SJ, McMurray JJ, Komajda M, McKelvie R, Baicu CF, Massie BM, Carson PE; I-PRESERVE Investigators. Prevalence and significance of alterations in cardiac structure and function in patients with heart failure and a preserved ejection fraction. Circulation. 2011 Dec 6;124(23):2491-501. doi: 10.1161/CIRCULATIONAHA.110.011031. Epub 2011 Nov 7. PMID 22064591
- [Derived] Krum H, Elsik M, Schneider HG, Ptaszynska A, Black M, Carson PE, Komajda M, Massie BM, McKelvie RS, McMurray JJ, Zile MR, Anand IS. Relation of peripheral collagen markers to death and hospitalization in patients with heart failure and preserved ejection fraction: results of the I-PRESERVE collagen substudy. Circ Heart Fail. 2011 Sep;4(5):561-8. doi: 10.1161/CIRCHEARTFAILURE.110.960716. Epub 2011 Jul 12. PMID 21750125
- [Derived] Anand IS, Rector TS, Cleland JG, Kuskowski M, McKelvie RS, Persson H, McMurray JJ, Zile MR, Komajda M, Massie BM, Carson PE. Prognostic value of baseline plasma amino-terminal pro-brain natriuretic peptide and its interactions with irbesartan treatment effects in patients with heart failure and preserved ejection fraction: findings from the I-PRESERVE trial. Circ Heart Fail. 2011 Sep;4(5):569-77. doi: 10.1161/CIRCHEARTFAILURE.111.962654. Epub 2011 Jun 29. PMID 21715583
- [Derived] Haass M, Kitzman DW, Anand IS, Miller A, Zile MR, Massie BM, Carson PE. Body mass index and adverse cardiovascular outcomes in heart failure patients with preserved ejection fraction: results from the Irbesartan in Heart Failure with Preserved Ejection Fraction (I-PRESERVE) trial. Circ Heart Fail. 2011 May;4(3):324-31. doi: 10.1161/CIRCHEARTFAILURE.110.959890. Epub 2011 Feb 24. PMID 21350053
- [Derived] Komajda M, Carson PE, Hetzel S, McKelvie R, McMurray J, Ptaszynska A, Zile MR, Demets D, Massie BM. Factors associated with outcome in heart failure with preserved ejection fraction: findings from the Irbesartan in Heart Failure with Preserved Ejection Fraction Study (I-PRESERVE). Circ Heart Fail. 2011 Jan;4(1):27-35. doi: 10.1161/CIRCHEARTFAILURE.109.932996. Epub 2010 Nov 10. PMID 21068341

RESULTS

PARTICIPANT FLOW:
Groups:
- Irbesartan; Placebo: titration from 75 to 300 mg, once daily (QD), up to 6 years
Period: Overall Study
Arm/Group | Irbesartan | Placebo
Started | 2067 (number randomized) | 2061 (number randomized)
Safety (Treated) Population | 2064 (Two participants were randomized but not treated; 1 randomized to irbesartan received placebo) | 2062 (One participant randomized to irbesartan received placebo.)
Completed | 1210 (completed double-blind therapy) | 1209 (completed double-blind therapy)
Not Completed | 857 | 852
Not completed — Lack of Efficacy | 9 | 9
Not completed — Adverse Event | 331 | 287
Not completed — Subject Withdrew Consent | 208 | 223
Not completed — Death | 154 | 170
Not completed — Lost to Follow-up | 19 | 24
Not completed — Noncompliance | 44 | 45
Not completed — No longer met study criteria | 4 | 5
Not completed — Study terminated by sponsor | 0 | 1
Not completed — Missing | 1 | 0
Not completed — Other Reasons | 87 | 88

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irbesartan | Placebo | Total
Number analyzed (Participants) | 2067 | 2061 | 4128
Age, Customized [Number; unit: participants]
  < 65 years | 376 | 364 | 740
  Between 65 and 74 years | 994 | 981 | 1975
  >=75 years | 697 | 716 | 1413
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (6.90) | 71.7 (7.00) | 71.6 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1227 | 1264 | 2491
  Male | 840 | 797 | 1637
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1934 | 1925 | 3859
  Black or African American | 39 | 43 | 82
  Asian | 19 | 15 | 34
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Other | 75 | 77 | 152
New York Heart Association (NYHA) Class [Number; unit: participants] — 1 participant in Placebo was not classified. NYHA Classes: I=No limitation of physical activity (does not cause undue fatigue, palpitation, or dyspnea). II=Slight limitation of physical activity (comfortable at rest, ordinary physical activity results in fatigue, palpitation, or dyspnea). III=Marked limitation of physical activity (comfortable at rest, less than ordinary activity causes fatigue, palpitation, or dyspnea). IV=Unable to carry out any physical activity without discomfort (symptoms of cardiac insufficiency at rest; discomfort is increased if any physical activity is undertaken).
  participants
    Class I (Mild) | 0 | 1 | 1
    Class II (Mild) | 426 | 444 | 870
    Class III (Moderate) | 1582 | 1562 | 3144
    Class IV (Severe) | 59 | 53 | 112
B-Type Natriuretic Peptide (Pro-BNP) [Geometric Mean (Inter-Quartile Range); unit: pg/mL] — Participant population=those participants with a baseline Pro-BNP measurement. Irbesartan (n=1765), Placebo (n=1798), Total (n=3563)
  pg/mL | 363.0 [140.0 to 994.0] | 345.2 [131.0 to 948.0] | 353.9 [135.0 to 974.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With First Occurrence of the Composite Outcome of Death (All Cause) or Protocol-Specified Cardiovascular (CV) Hospitalization at Given Timepoints
Description: Treatment comparisons for time to first occurrence of composite outcome of all-cause death (composite outcome of death) or protocol-specified CV hospitalization. Protocol-specified CV hospitalizations include those ≥24 hrs or involving a calendar date change for a primary cause of worsening heart failure, unstable angina, myocardial infarction, ventricular or atrial dysrhythmia, or stroke, that also require intravenous or intramuscular therapy or a related procedure or significant augmentation of oral therapy. In addition, MI or stroke during any hospitalization are included.
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: Randomized Participants
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage at 1 Year | 12.3 | 12.1
  Percentage at 2 Years | 20.7 | 21.3
  Percentage at 3 Years | 26.4 | 28.4
  Percentage at 4 Years | 32.9 | 34.2
  Percentage at 5 Years | 39.2 | 39.5

2. Secondary Outcome: Percentage of Participants Experiencing Heart Failure Mortality or Heart Failure Hospitalization at Given Time Points
Description: Treatment comparisons for time to heart failure mortality or heart failure hospitalization
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: Randomized Participants
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage at 1 Year | 7.9 | 8.2
  Percentage at 2 Years | 12.9 | 13.7
  Percentage at 3 Years | 15.7 | 17.2
  Percentage at 4 Years | 19.8 | 20.3
  Percentage at 5 Years | 23.6 | 23.8

3. Secondary Outcome: Minnesota Living With Heart Failure (MLwHF) Total Score (Sum of Questions 1-21) at Month 6 and Month 14
Description: Mean score and adjusted mean change from baseline in Minnesota Living with Heart Failure (MLWHF) questionnaire, a 21-item, patient-reported, 6-point (ranging from 0-5; higher score=poorer quality of life; highest possible score=105) measurement of quality of life in persons with heart failure.
Time Frame: Baseline, Month 6, Month 14
Population: Participants with baseline score and score at timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo - Month 6: Cohort of participants in Placebo group with MLwHF scores at Baseline and Month 6
- Irbesartan - Month 6: Cohort of participants in Irbesartan group with MLwHF scores at Baseline and Month 6
- Placebo - Month 14: Cohort of participants in Placebo group with MLwHF scores at Baseline and Month 14
- Irbesartan - Month 14: Cohort of participants in Irbesartan group with MLwHF scores at Baseline and Month 14
Arm/Group | Placebo - Month 6 | Irbesartan - Month 6 | Placebo - Month 14 | Irbesartan - Month 14
Number analyzed (Participants) | 1552 | 1550 | 1434 | 1428
units on a scale
  Baseline Mean Score | 42.7 (0.52) | 43.0 (0.53) | 42.7 (0.53) | 42.8 (0.55)
  Mean Score at Timepoint | 32.9 (0.48) | 33.2 (0.50) | 31.6 (0.50) | 32.1 (0.50)
  Adjusted Mean Change from Baseline | -10.0 (0.41) | -9.8 (0.41) | -11.2 (0.42) | -10.6 (0.42)
Statistical Analysis 1: Comparison: Placebo - Month 6 vs Irbesartan - Month 6; Comparison of 2 treatment arms at Month 6 (first 2 columns); Test type: Superiority or Other; Mixed Models Analysis; baseline score used as covariate; treatment, visit, treatment-by-visit, & baseline angiotensin-converting enzyme (ACE) inhibitors used as predictors; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.8 to 1.3]
Statistical Analysis 2: Comparison: Placebo - Month 14 vs Irbesartan - Month 14; comparison of 2 treatment arms at Month 14 (columns 3 and 4); Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.5 to 1.7]

4. Secondary Outcome: Minnesota Living With Heart Failure (MLwHF) Total Score (Sum of Questions 1-21) at Final Visit
Description: Mean score at baseline and final visit in Minnesota Living with Heart Failure (MLWHF) questionnaire, a 21-item, patient-reported, 6-point (ranging from 0-5; higher score=poorer quality of life; highest possible score=105) measurement of quality of life in persons with heart failure.
Time Frame: Baseline, Final Visit=last scheduled visit specified in the protocol at conclusion of the entire study by the sponsor. The trial was designed to end after 1440 primary endpoint events, projected duration=6.0 ± 0.5 years.
Population: Participants with baseline score and score at timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo - Final Visit: Cohort of participants in Placebo group with MLwHF scores at Baseline and Final Visit
- Irbesartan - Final Visit: Cohort of participants in Irbesartan group with MLwHF scores at Baseline and Final Visit
Arm/Group | Placebo - Final Visit | Irbesartan - Final Visit
Number analyzed (Participants) | 2067 | 2061
units on a scale
  Baseline Mean | 42.5 (0.49) | 38.9 (0.67)
  Final Visit Mean | 42.6 (0.51) | 38.3 (0.69)

5. Secondary Outcome: Change From Baseline in B-Type Natriuretic Peptide (Pro-BNP) at Month 6 and Month 14
Description: Adjusted ratio to baseline in geometric mean in Pro-BNP in the blood. Ratio to Baseline = On-therapy geometric mean divided by baseline geometric mean. A lower score signifies improvement. Change from baseline adjusted for baseline value and angiotensin converting enzyme inhibitor use at baseline. Analysis uses natural logarithms of excretion rate values.
Time Frame: Baseline, Month 6, Month 14
Population: number of participants with measurement at baseline and at timepoint
Measure: Geometric Mean (Standard Error); unit: pg/mL
Groups:
- Placebo - Month 6: Placebo cohort with measurements at baseline and Month 6.
- Irbesartan - Month 6: Irbesartan cohort with measurements at Baseline and Month 6.
- Placebo - Month 14: Placebo cohort with measurements at Baseline and Month 14.
- Irbesartan - Month 14: Irbesartan cohort with measurements at Baseline and Month 14.
Arm/Group | Placebo - Month 6 | Irbesartan - Month 6 | Placebo - Month 14 | Irbesartan - Month 14
Number analyzed (Participants) | 1336 | 1337 | 1295 | 1281
pg/mL | 0.98 (0.023) | 0.93 (0.022) | 1.00 (0.026) | 1.01 (0.026)

6. Secondary Outcome: Percentage of Participants Experiencing CV Death, Non-Fatal Myocardial Infarction (MI), or Non-Fatal Stroke at Given Timepoints
Description: Treatment comparisons for time to cardiovascular death, non-fatal MI, or non-fatal stroke.
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: Randomized Participants
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage at 1 Year | 5.2 | 4.2
  Percentage at 2 Years | 8.7 | 9.3
  Percentage at 3 Years | 12.9 | 13.6
  Percentage at 4 Years | 17.2 | 17.6
  Percentage at 5 Years | 23.0 | 22.4

7. Secondary Outcome: Percentage of Participants Experiencing Cardiovascular Death at Given Timepoints
Description: Treatment comparisons for time to cardiovascular death
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: Randomized Subjects
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage 1 Year | 3.3 | 3.0
  Percentage 2 Years | 6.2 | 6.5
  Percentage 3 Years | 9.6 | 10.0
  Percentage at 4 Years | 13.0 | 13.1
  Percentage at 5 Years | 18.0 | 17.1

8. Secondary Outcome: Percentage of Participants Experiencing All-cause Death at Given Time Points
Description: Treatment comparisons for time to all-cause death
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: Randomized subjects
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage at 1 Year | 4.1 | 3.8
  Percentage at 2 Years | 8.1 | 8.6
  Percentage at 3 Years | 12.8 | 13.8
  Percentage at 4 Years | 17.9 | 18.5
  Percentage at 5 Years | 25.0 | 23.6

9. Secondary Outcome: Change From Baseline in the New York Heart Association (NYHA) Functional Class at Month 6, Month 10, Month 14, and Final Visit
Description: NYHA functional classification=4-tiered system relating symptoms to everyday activities & quality of life. (See Reporting Groups for description of each class.) Change of NYHA functional class from baseline was grouped into 3 categories: improved, unchanged, or worsened (based on case report form [CRF] assessment). If a post-randomization CRF assessment was missing or participant died, was hospitalized for worsening heart failure or discontinued study medication for worsening heart failure, the participant was classified as Major Event.
Time Frame: Baseline, Month 6, Month 10, Month 14, Final Visit. The trial was designed to end after 1440 primary endpoint events, projected duration=6.0 ± 0.5 years.
Population: Randomized participants with measurement at baseline and Month 6, Month 10, Month 14, and Final Visit
Measure: Number; unit: participants
Groups:
- Irbesartan Baseline Class I or II: Class I (Mild): No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath). Class II (Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
- Irbesartan Class III or IV: Class III (Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV (Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased.
Arm/Group | Irbesartan Baseline Class I or II | Irbesartan Class III or IV | Irbesartan Baseline All Classes Combined | Placebo Baseline Class I or II | Placebo Class III or IV | Placebo Baseline All Classes Combined
Number analyzed (Participants) | 426 | 1641 | 2067 | 445 | 1615 | 2060
participants
  Month 6 - Improved | 55 | 881 | 936 | 47 | 834 | 881
  Month 6 - Unchanged | 310 | 656 | 966 | 338 | 678 | 1016
  Month 6 - Worsened | 41 | 7 | 48 | 47 | 4 | 51
  Month 6 - Major Event | 2 | 8 | 10 | 2 | 12 | 14
  Month 6 - No Data | 18 | 89 | 107 | 11 | 87 | 98
  Month 10 - Improved | 44 | 904 | 948 | 42 | 860 | 902
  Month 10 - Unchanged | 294 | 617 | 911 | 317 | 622 | 939
  Month 10 - Worsened | 53 | 5 | 58 | 63 | 8 | 71
  Month 10 - Major Event | 10 | 31 | 41 | 9 | 33 | 42
  Month 10 - No Data | 25 | 84 | 109 | 14 | 92 | 106
  Month 14 - Improved | 38 | 895 | 933 | 39 | 863 | 902
  Month 14 - Unchanged | 287 | 579 | 866 | 312 | 578 | 890
  Month 14 - Worsened | 50 | 11 | 61 | 62 | 7 | 69
  Month 14 - Major Event | 22 | 53 | 75 | 16 | 64 | 80
  Month 14 - No Data | 29 | 103 | 132 | 16 | 103 | 119
  Final Visit - Improved | 42 | 886 | 928 | 42 | 840 | 882
  Final Visit - Unchanged | 230 | 428 | 658 | 254 | 440 | 694
  Final Visit - Worsened | 68 | 29 | 97 | 78 | 29 | 107
  Final Visit - Major Event | 75 | 249 | 324 | 66 | 254 | 320
  Final Visit - No Data | 11 | 49 | 60 | 5 | 52 | 57

10. Secondary Outcome: Physician Assessment of Heart Failure Status at Month 6, Month 14, and Final Visit Compared With Baseline
Description: This was an assessment of the change in overall physician opinion of change from baseline status. Assessments are directly based on the Case Report Form (CRF). If the post-randomization CRF assessment was missing and the subject died, was hospitalized for worsening heart failure, or discontinued study medication for worsening heart failure, the subject was considered as having a Major Event. Participants who are summarized under Major Events are categorized as Worsened Markedly.
Time Frame: Baseline, Month 6, Month 14, Final Visit. The trial was designed to end after 1440 primary endpoint events, projected duration=6.0 ± 0.5 years.
Measure: Number; unit: participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
participants
  Month 6 - Improved Markedly | 230 | 198
  Month 6 - Improved Moderately | 562 | 575
  Month 6 - Improved Slightly | 533 | 529
  Month 6 - Unchanged | 528 | 541
  Month 6 - Worsened Slightly | 60 | 58
  Month 6 - Worsened Moderately | 17 | 16
  Month 6 - Worsened Markedly | 0 | 4
  Month 6 - Major Event | 8 | 8
  Month 6 - No Data | 129 | 132
  Month 14 - Improved Markedly | 214 | 195
  Month 14 - Improved Moderately | 546 | 537
  Month 14 - Improved Slightly | 442 | 435
  Month 14 - Unchanged | 507 | 548
  Month 14 - Worsened Slightly | 72 | 73
  Month 14 - Worsened Moderately | 21 | 19
  Month 14 - Worsened Markedly | 5 | 6
  Month 14 - Major Event | 75 | 79
  Month 14 - No Data | 185 | 169
  Final Visit - Improved Markedly | 180 | 186
  Final Visit - Improved Moderately | 430 | 367
  Final Visit - Improved Slightly | 344 | 361
  Final Visit - Unchanged | 477 | 504
  Final Visit - Worsened Slightly | 117 | 117
  Final Visit - Worsened Moderately | 41 | 56
  Final Visit - Worsened Markedly | 23 | 28
  Final Visit - Major Event | 364 | 350
  Final Visit - No Data | 91 | 92

11. Secondary Outcome: Participant Assessment of Heart Failure Status at Month 6, Month 14, and Final Visit Compared With Baseline
Description: Assessments are directly based on the Case Report Form (CRF). If the post-randomization CRF assessment was missing and the subject died, was hospitalized for worsening heart failure, or discontinued study medication for worsening heart failure, the subject was considered as having a Major Event. Participants who are summarized under Major Events are categorized as Worsened Markedly.
Time Frame: as for outcome 10
Population: Randomized Participants
Measure: Number; unit: Participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
Participants
  Month 6 - Improved Markedly | 235 | 230
  Month 6 - Improved Moderately | 552 | 563
  Month 6 - Improved Slightly | 529 | 519
  Month 6 - Unchanged | 537 | 529
  Month 6 - Worsened Slightly | 63 | 69
  Month 6 - Worsened Moderately | 13 | 20
  Month 6 - Worsened Markedly | 8 | 8
  Month 6 - Major Event | 8 | 7
  Month 6 - No Data | 122 | 116
  Month 14 - Improved Markedly | 234 | 206
  Month 14 - Improved Moderately | 532 | 534
  Month 14 - Improved Slightly | 461 | 450
  Month 14 - Unchanged | 503 | 527
  Month 14 - Worsened Slightly | 78 | 82
  Month 14 - Worsened Moderately | 30 | 35
  Month 14 - Worsened Markedly | 8 | 7
  Month 14 - Major Event | 68 | 74
  Month 14 - No Data | 153 | 146
  Final Visit - Improved Markedly | 207 | 201
  Final Visit - Improved Moderately | 378 | 339
  Final Visit - Improved Slightly | 332 | 352
  Final Visit - Unchanged | 480 | 495
  Final Visit - Worsened Slightly | 121 | 109
  Final Visit - Worsened Moderately | 52 | 76
  Final Visit - Worsened Markedly | 25 | 28
  Final Visit - Major Event | 396 | 383
  Final Event - No Data | 76 | 78

12. Secondary Outcome: Participant Assessment of Fatigue at Month 6, Month 14, and Final Visit Compared With Baseline
Description: as for outcome 11
Time Frame: as for outcome 10
Population: Randomized Participants
Measure: Number; unit: Participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
Participants
  Month 6 - Improved Markedly | 193 | 200
  Month 6 - Improved Moderately | 523 | 519
  Month 6 - Improved Slightly | 504 | 471
  Month 6 - Unchanged | 579 | 596
  Month 6 - Worsened Slightly | 97 | 101
  Month 6 - Worsened Moderately | 28 | 38
  Month 6 - Worsened Markedly | 13 | 13
  Month 6 - Major Event | 8 | 7
  Month 6 - No Data | 122 | 116
  Month 14 - Improved Markedly | 195 | 182
  Month 14 - Improved Moderately | 513 | 489
  Month 14 - Improved Slightly | 439 | 443
  Month 14 - Unchanged | 525 | 559
  Month 14 - Worsened Slightly | 115 | 109
  Month 14 - Worsened Moderately | 48 | 43
  Month 14 - Worsened Markedly | 11 | 16
  Month 14 - Major Event | 68 | 74
  Month 14 - No Data | 153 | 146
  Final Visit - Improved Markedly | 157 | 178
  Final Visit - Improved Moderately | 361 | 300
  Final Visit - Improved Slightly | 319 | 337
  Final Visit - Unchanged | 479 | 477
  Final Visit - Worsened Slightly | 166 | 176
  Final Visit - Worsened Moderately | 80 | 90
  Final Visit - Worsened Markedly | 34 | 42
  Final Visit - Major Event | 395 | 383
  Final Visit - No Data | 76 | 78

13. Secondary Outcome: Participant Assessment of Dyspnea at Month 6, Month 14, and Final Visit Compared With Baseline
Description: as for outcome 11
Time Frame: as for outcome 10
Population: Randomized Participants
Measure: Number; unit: Participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
Participants
  Month 6 - Improved Markedly | 255 | 276
  Month 6 - Improved Moderately | 549 | 536
  Month 6 - Improved Slightly | 512 | 501
  Month 6 - Unchanged | 508 | 510
  Month 6 - Worsened Slightly | 83 | 83
  Month 6 - Worsened Moderately | 22 | 22
  Month 6 - Worsened Markedly | 9 | 10
  Month 6 - Major Event | 8 | 7
  Month 6 - No Data | 121 | 116
  Month 14 - Improved Markedly | 247 | 232
  Month 14 - Improved Moderately | 519 | 531
  Month 14 - Improved Slightly | 460 | 430
  Month 14 - Unchanged | 476 | 509
  Month 14 - Worsened Slightly | 103 | 90
  Month 14 - Worsened Moderately | 28 | 39
  Month 14 - Worsened Markedly | 13 | 10
  Month 14 - Major Event | 68 | 74
  Month 14 - No Data | 153 | 146
  Final Visit - Improved Markedly | 213 | 212
  Final Visit - Improved Moderately | 382 | 339
  Final Visit - Improved Slightly | 328 | 335
  Final Visit - Unchanged | 460 | 461
  Final Visit - Worsened Slightly | 114 | 145
  Final Visit - Worsened Moderately | 64 | 75
  Final Visit - Worsened Markedly | 35 | 32
  Final Visit - Major Event | 395 | 384
  Final Visit - No Data | 76 | 78

14. Secondary Outcome: Percentage of Participants Experiencing CV Death or CV Hospitalization at Given Timepoints
Description: Treatment comparisons for time to CV death or CV hospitalization. Protocol-specified CV hospitalizations include hospitalizations ≥24 hrs or involve a calendar date change for a primary cause of worsening heart failure, unstable angina, myocardial infarction, ventricular dysrhythmia, atrial dysrhythmia or stroke that also requires intravenous or intramuscular therapy or a related procedure or significant augmentation of oral therapy. Protocol specified CV hospitalizations also include myocardial infarction or stroke occurring during any hospitalization.
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage at 1 Year | 11.6 | 11.4
  Percentage at 2 Years | 19.2 | 20.0
  Percentage at 3 Years | 24.2 | 25.8
  Percentage at 4 Years | 30.0 | 30.9
  Percentage at 5 Years | 35.0 | 35.8

15. Secondary Outcome: Percentage of Participants Experiencing Protocol-specified Cardiovascular (CV) Hospitalization at Given Timepoints
Description: Treatment comparisons for time to protocol-specified CV hospitalization. Protocol-specified CV hospitalizations include hospitalizations ≥24 hrs or involve a calendar date change for a primary cause of worsening heart failure, unstable angina, myocardial infarction, ventricular dysrhythmia, atrial dysrhythmia or stroke that also requires intravenous or intramuscular therapy or a related procedure or significant augmentation of oral therapy. Protocol specified CV hospitalizations also include myocardial infarction or stroke occurring during any hospitalization.
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 2067 | 2061
percentage of participants
  Percentage at 1 Year | 9.7 | 9.8
  Percentage at 2 Years | 16.3 | 17.1
  Percentage at 3 Years | 20.5 | 21.7
  Percentage at 4 Years | 24.8 | 25.9
  Percentage at 5 Years | 28.5 | 29.0

16. Secondary Outcome: Percentage of Participants With New Onset of Diabetes Among Subjects With No Prior Diabetes History at Given Timepoints
Description: Treatment comparisons for time to new onset of diabetes (from adverse event reporting) among subjects with no prior history of diabetes.
Time Frame: Year 1, Year 2, Year 3, Year 4, Year 5
Population: Randomized participants with no prior diabetes history
Measure: Number; unit: percentage of participants
Arm/Group | Irbesartan | Placebo
Number analyzed (Participants) | 1495 | 1496
percentage of participants
  Percentage at 1 Year | 0.7 | 1.2
  Percentage at 2 Years | 2.1 | 2.8
  Percentage at 3 Years | 3.1 | 3.9
  Percentage at 4 Years | 4.6 | 5.4
  Percentage at 5 Years | 5.2 | 6.2

17. Secondary Outcome: Mean Change From Baseline in Glomerular Filtration Rate (GFR) at Month 6, Month 18, and Month 30
Description: Based on the Cockcroft-Gault formula calculation, a commonly used surrogate marker to estimate creatinine clearance, which in turn is an approximate measure of GFR. It employs serum creatinine measurements and a patient's weight to predict the creatinine clearance. Adjusted for baseline GFR and angiotensin-converting enzyme inhibitor use at baseline (ACE-I). A decrease from baseline signifies worsening. The adjusted mean change from baseline value is from the model (calculated prior to rounding), whereas the other two points are the baseline mean and post mean.
Time Frame: Baseline, Month 6, Month 18, Month 30
Population: Participants with baseline score and score at timepoint.
Measure: Mean (Standard Error); unit: mL/min/1.73m2
Groups:
- Placebo - Month 6: Cohort of participants in Placebo group with GFR assessment at Baseline and Month 6
- Irbesartan - Month 6: Cohort of participants in irbesartan group with GFR assessment at Baseline and Month 6
- Placebo - Month 18: Cohort of participants in Placebo group with GFR assessment at Baseline and Month 18
- Irbesartan - Month 18: Cohort of participants in irbesartan group with GFR assessment at Baseline and Month 18
- Placebo - Month 30: Cohort of participants in Placebo group with GFR assessment at Baseline and Month 30
- Irbesartan - Month 30: Cohort of participants in irbesartan group with GFR assessment at Baseline and Month 30
Arm/Group | Placebo - Month 6 | Irbesartan - Month 6 | Placebo - Month 18 | Irbesartan - Month 18 | Placebo - Month 30 | Irbesartan - Month 30
Number analyzed (Participants) | 1741 | 1734 | 1406 | 1379 | 1270 | 1225
mL/min/1.73m2
  Baseline Mean | 73.02 (0.536) | 73.13 (0.538) | 73.58 (0.589) | 73.49 (0.591) | 73.34 (0.606) | 74.37 (0.630)
  Post-Baseline Mean | 71.97 (0.527) | 69.21 (0.562) | 70.88 (0.583) | 68.00 (0.596) | 69.51 (0.589) | 67.05 (0.595)
  Adjusted Mean Change | -1.07 (0.393) | -3.91 (0.394) | -2.69 (0.436) | -5.50 (0.440) | -4.02 (0.442) | -7.12 (0.450)

18. Secondary Outcome: Mean Change From Baseline in Glomerular Filtration Rate (GFR)at Month 42, Month 54, Month 66
Description: as for outcome 17
Time Frame: Baseline, Month 42, Month 54, Month 66
Population: Participants with baseline score and score at timepoint.
Measure: Mean (Standard Error); unit: mL/min/1.73m2
Groups:
- Placebo - Month 42: Cohort of participants in Placebo group with GFR assessment at Baseline and Month 42
- Irbesartan - Month 42: Cohort of participants in irbesartan group with GFR assessment at Baseline and Month 42
- Placebo - Month 54; Irbesartan - Month 54: Cohort of participants in Placebo group with GFR assessment at Baseline and Month 54
- Placebo - Month 66: Cohort of participants in Placebo group with GFR assessment at Baseline and Month 66
- Irbesartan - Month 66: Cohort of participants in irbesartan group with GFR assessment at Baseline and Month 66
Arm/Group | Placebo - Month 42 | Irbesartan - Month 42 | Placebo - Month 54 | Irbesartan - Month 54 | Placebo - Month 66 | Irbesartan - Month 66
Number analyzed (Participants) | 928 | 921 | 429 | 455 | 22 | 22
mL/min/1.73m2
  Baseline Mean | 74.37 (0.715) | 74.95 (0.711) | 75.29 (1.075) | 75.17 (1.052) | 63.47 (5.596) | 71.84 (5.919)
  Post-Baseline Mean | 71.34 (0.700) | 67.48 (0.715) | 72.65 (1.048) | 68.24 (1.055) | 60.09 (5.832) | 64.85 (6.301)
  Adjusted Mean Change | -3.14 (0.559) | -7.36 (0.561) | -2.63 (0.863) | -6.93 (0.838) | -4.91 (4.534) | -5.46 (4.534)

19. Secondary Outcome: Number of Participants With New Onset Atrial Fibrillation (AF) Among Those With No Prior AF History or Evidence of AF on Baseline Electrocardiograph (ECG)
Description: Frequency of new onset AF in participants with no prior AF history or evidence of AF on baseline ECG. Stratified by use of angiotensin-converting enzyme (ACE) inhibitors and measured by adverse events reporting and final ECG recording read by the investigator.
Time Frame: Baseline, Final Visit
Population: Randomized subjects (total=4128) with no prior AF history or evidence of AF on baseline ECG, stratified by use of ACE-I
Measure: Number; unit: participants
Arm/Group | Irbesartan + ACE-I Use | Placebo + ACE-I Use | Irbesartan no ACE-I Use | Placebo no ACE-I Use
Number analyzed (Participants) | 538 | 510 | 1529 | 1551
participants
  No prior AF history or Evidence on Baseline ECG | 366 | 344 | 1089 | 1102
  Participants with New Onset Atrial Fibrillation | 35 | 29 | 103 | 99

ADVERSE EVENTS:
Time Frame: SAEs: from start of study through last treatment +30 days; AEs: through the last dose +1 day.
Arm/Group | IRBESARTAN | PLACEBO
Serious Adverse Events (participants affected / at risk) | 1146/2064 | 1155/2062
Other Adverse Events (participants affected / at risk) | 1255/2064 | 1191/2062
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IRBESARTAN (N=2064) | PLACEBO (N=2062)
CATARACT (Eye disorders) | 16 | 10
DIPLOPIA (Eye disorders) | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 3
MACULOPATHY (Eye disorders) | 0 | 2
RETINOPATHY (Eye disorders) | 0 | 1
IRIDOCYCLITIS (Eye disorders) | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 2
MACULAR RUPTURE (Eye disorders) | 0 | 1
ATROPHY OF GLOBE (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 2 | 1
BLINDNESS UNILATERAL (Eye disorders) | 1 | 0
CORNEAL DEGENERATION (Eye disorders) | 0 | 1
DIABETIC RETINOPATHY (Eye disorders) | 1 | 1
MACULAR DEGENERATION (Eye disorders) | 0 | 1
ULCERATIVE KERATITIS (Eye disorders) | 1 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 1 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 0
RETINAL VEIN OCCLUSION (Eye disorders) | 1 | 0
RETINAL ARTERY EMBOLISM (Eye disorders) | 1 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 | 0
ANGIOGRAM (Investigations) | 0 | 1
WEIGHT DECREASED (Investigations) | 2 | 4
TROPONIN INCREASED (Investigations) | 0 | 1
BLOOD URINE PRESENT (Investigations) | 0 | 1
BLOOD UREA INCREASED (Investigations) | 0 | 1
CHEST X-RAY ABNORMAL (Investigations) | 0 | 1
HAEMOGLOBIN ABNORMAL (Investigations) | 1 | 0
HEART RATE INCREASED (Investigations) | 0 | 2
BLOOD GLUCOSE ABNORMAL (Investigations) | 1 | 0
BLOOD ALCOHOL INCREASED (Investigations) | 0 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 3
BLOOD PRESSURE INCREASED (Investigations) | 4 | 5
ELECTROCARDIOGRAM CHANGE (Investigations) | 0 | 2
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 1
BLOOD POTASSIUM INCREASED (Investigations) | 1 | 1
BLOOD CREATININE INCREASED (Investigations) | 1 | 2
COAGULATION TIME PROLONGED (Investigations) | 0 | 1
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 1 | 0
RESPIRATORY RATE DECREASED (Investigations) | 1 | 0
CARCINOEMBRYONIC ANTIGEN INCREASED (Investigations) | 0 | 1
SCAN MYOCARDIAL PERFUSION ABNORMAL (Investigations) | 1 | 0
BLOOD PRESSURE ORTHOSTATIC ABNORMAL (Investigations) | 0 | 1
PULMONARY ARTERIAL PRESSURE INCREASED (Investigations) | 1 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 2 | 4
ARRHYTHMIA (Cardiac disorders) | 15 | 11
BRADYCARDIA (Cardiac disorders) | 14 | 13
TACHYCARDIA (Cardiac disorders) | 10 | 4
PALPITATIONS (Cardiac disorders) | 2 | 5
PERICARDITIS (Cardiac disorders) | 0 | 3
SINUS ARREST (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 15 | 11
CARDIAC ARREST (Cardiac disorders) | 9 | 9
CARDIAC ASTHMA (Cardiac disorders) | 2 | 7
ANGINA PECTORIS (Cardiac disorders) | 59 | 61
ANGINA UNSTABLE (Cardiac disorders) | 86 | 78
BRADYARRHYTHMIA (Cardiac disorders) | 2 | 2
CARDIAC FAILURE (Cardiac disorders) | 274 | 275
TACHYARRHYTHMIA (Cardiac disorders) | 2 | 2
CARDIAC DISORDER (Cardiac disorders) | 3 | 1
NODAL ARRHYTHMIA (Cardiac disorders) | 1 | 2
SINOATRIAL BLOCK (Cardiac disorders) | 0 | 2
SINUS ARRHYTHMIA (Cardiac disorders) | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 5 | 6
SINUS BRADYCARDIA (Cardiac disorders) | 5 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
ATRIAL TACHYCARDIA (Cardiac disorders) | 2 | 0
BIFASCICULAR BLOCK (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 105 | 104
BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 | 1
CARDIAC HYPERTROPHY (Cardiac disorders) | 1 | 0
CONDUCTION DISORDER (Cardiac disorders) | 1 | 0
DRESSLER'S SYNDROME (Cardiac disorders) | 0 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 5 | 15
AORTIC VALVE DISEASE (Cardiac disorders) | 1 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 12 | 10
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
ADAMS-STOKES SYNDROME (Cardiac disorders) | 0 | 1
AORTIC VALVE STENOSIS (Cardiac disorders) | 6 | 2
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 5 | 2
CARDIAC VALVE DISEASE (Cardiac disorders) | 0 | 1
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 | 1
MITRAL VALVE PROLAPSE (Cardiac disorders) | 0 | 1
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 42 | 47
PAROXYSMAL ARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 2 | 7
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 15 | 14
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 2 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 16 | 15
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 | 0
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 8 | 10
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 2
CHORDAE TENDINAE RUPTURE (Cardiac disorders) | 1 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 5 | 2
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 0 | 1
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 3 | 6
VENTRICULAR FIBRILLATION (Cardiac disorders) | 2 | 6
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 | 1
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 5 | 7
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 2
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 3 | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 3 | 2
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 55 | 61
CORONARY ARTERY DISSECTION (Cardiac disorders) | 1 | 0
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 39 | 33
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 | 1
SILENT MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 5 | 10
CARDIOVASCULAR DECONDITIONING (Cardiac disorders) | 1 | 0
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 3 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 11 | 8
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 3 | 0
SUPRAVENTRICULAR TACHYARRHYTHMIA (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 4
SHOCK (Vascular disorders) | 1 | 2
EMBOLISM (Vascular disorders) | 2 | 2
ARTERITIS (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 6 | 3
ISCHAEMIA (Vascular disorders) | 1 | 6
PHLEBITIS (Vascular disorders) | 1 | 2
INFARCTION (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 2 | 2
HAEMORRHAGE (Vascular disorders) | 2 | 1
HYPOTENSION (Vascular disorders) | 25 | 20
HYPERTENSION (Vascular disorders) | 33 | 35
VARICOSE VEIN (Vascular disorders) | 2 | 4
ANGIOSCLEROSIS (Vascular disorders) | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 4 | 3
AORTIC STENOSIS (Vascular disorders) | 5 | 5
ARTERIAL RUPTURE (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 3 | 1
THROMBOPHLEBITIS (Vascular disorders) | 1 | 1
ANEURYSM RUPTURED (Vascular disorders) | 0 | 2
VENOUS THROMBOSIS (Vascular disorders) | 1 | 2
EXTREMITY NECROSIS (Vascular disorders) | 1 | 0
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 | 3
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 | 0
TEMPORAL ARTERITIS (Vascular disorders) | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 10 | 8
PERIPHERAL EMBOLISM (Vascular disorders) | 5 | 2
VARICOSE ULCERATION (Vascular disorders) | 1 | 0
ARTERIAL HAEMORRHAGE (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 7 | 4
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 3
PERIPHERAL ISCHAEMIA (Vascular disorders) | 7 | 4
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 | 1
ARTERIAL INSUFFICIENCY (Vascular disorders) | 0 | 1
ARTERIAL STENOSIS LIMB (Vascular disorders) | 0 | 3
ESSENTIAL HYPERTENSION (Vascular disorders) | 0 | 1
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1 | 0
VASCULAR INSUFFICIENCY (Vascular disorders) | 2 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 3 | 4
VASCULAR PSEUDOANEURYSM (Vascular disorders) | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 4 | 1
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 5 | 4
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 1
DIABETIC VASCULAR DISORDER (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS OBLITERANS (Vascular disorders) | 2 | 3
VISCERAL ARTERIAL ISCHAEMIA (Vascular disorders) | 0 | 1
CARDIOVASCULAR INSUFFICIENCY (Vascular disorders) | 0 | 1
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 5 | 3
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 2
GOITRE (Endocrine disorders) | 3 | 5
THYROIDITIS (Endocrine disorders) | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 3 | 1
HYPERTHYROIDISM (Endocrine disorders) | 2 | 1
THYROID DISORDER (Endocrine disorders) | 0 | 1
BASEDOW'S DISEASE (Endocrine disorders) | 1 | 0
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 1
SOPOR (Psychiatric disorders) | 1 | 0
STRESS (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 3 | 2
DELIRIUM (Psychiatric disorders) | 1 | 1
AGITATION (Psychiatric disorders) | 0 | 1
ALCOHOLISM (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 9 | 6
NERVOUSNESS (Psychiatric disorders) | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 1
DISORIENTATION (Psychiatric disorders) | 2 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 1
DRUG DEPENDENCE (Psychiatric disorders) | 1 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 3 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 7 | 3
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 | 0
DYSTHYMIC DISORDER (Psychiatric disorders) | 1 | 0
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 | 1
PERSONALITY DISORDER (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
SOCIAL AVOIDANT BEHAVIOUR (Psychiatric disorders) | 0 | 1
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 | 1
OBSESSIVE-COMPULSIVE DISORDER (Psychiatric disorders) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 3
HEPATITIS (Hepatobiliary disorders) | 0 | 2
CHOLANGITIS (Hepatobiliary disorders) | 1 | 2
CHOLESTASIS (Hepatobiliary disorders) | 1 | 1
BILIARY COLIC (Hepatobiliary disorders) | 2 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 12 | 8
CHOLELITHIASIS (Hepatobiliary disorders) | 21 | 25
LIVER DISORDER (Hepatobiliary disorders) | 1 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 4
BILIARY FISTULA (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 2
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 | 0
HYDROCHOLECYSTIS (Hepatobiliary disorders) | 1 | 0
CARDIAC CIRRHOSIS (Hepatobiliary disorders) | 0 | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 3 | 3
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 5 | 3
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 4 | 2
HEPATITIS CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
AMPULLA OF VATER STENOSIS (Hepatobiliary disorders) | 0 | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
AMYLOIDOSIS (Immune system disorders) | 0 | 1
SARCOIDOSIS (Immune system disorders) | 0 | 1
IODINE ALLERGY (Immune system disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 2
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
COMA (Nervous system disorders) | 0 | 1
TREMOR (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 36 | 41
DEMENTIA (Nervous system disorders) | 0 | 3
EPILEPSY (Nervous system disorders) | 2 | 1
HEADACHE (Nervous system disorders) | 1 | 5
SCIATICA (Nervous system disorders) | 3 | 2
DIZZINESS (Nervous system disorders) | 9 | 12
HYPOTONIA (Nervous system disorders) | 0 | 1
NEURALGIA (Nervous system disorders) | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 4
DYSARTHRIA (Nervous system disorders) | 1 | 0
HEMIPLEGIA (Nervous system disorders) | 0 | 2
HYPERTONIA (Nervous system disorders) | 3 | 1
MONOPLEGIA (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 5 | 4
SOMNOLENCE (Nervous system disorders) | 0 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 2
MONOPARESIS (Nervous system disorders) | 1 | 0
BRAIN INJURY (Nervous system disorders) | 2 | 0
DROP ATTACKS (Nervous system disorders) | 0 | 1
DYSAESTHESIA (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 2
SENSORY LOSS (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 3 | 3
FACIAL PARESIS (Nervous system disorders) | 1 | 1
GLOBAL AMNESIA (Nervous system disorders) | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 1 | 0
BALANCE DISORDER (Nervous system disorders) | 2 | 0
CEREBROSCLEROSIS (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 14 | 25
PARTIAL SEIZURES (Nervous system disorders) | 1 | 0
SPINAL HAEMATOMA (Nervous system disorders) | 1 | 0
MENTAL IMPAIRMENT (Nervous system disorders) | 2 | 1
MOTOR DYSFUNCTION (Nervous system disorders) | 1 | 0
MYASTHENIA GRAVIS (Nervous system disorders) | 0 | 1
SYNCOPE VASOVAGAL (Nervous system disorders) | 2 | 0
VASCULAR DEMENTIA (Nervous system disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 5 | 2
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 | 0
RADICULAR SYNDROME (Nervous system disorders) | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 3 | 2
DIABETIC NEUROPATHY (Nervous system disorders) | 0 | 3
HAEMORRHAGIC STROKE (Nervous system disorders) | 5 | 4
PARKINSON'S DISEASE (Nervous system disorders) | 1 | 1
SPINAL CLAUDICATION (Nervous system disorders) | 1 | 0
WALLENBERG SYNDROME (Nervous system disorders) | 1 | 0
CEREBELLAR HAEMATOMA (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 2
GRAND MAL CONVULSION (Nervous system disorders) | 1 | 0
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
COORDINATION ABNORMAL (Nervous system disorders) | 1 | 0
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 3 | 2
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 2 | 2
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 7 | 5
SPINAL CORD COMPRESSION (Nervous system disorders) | 3 | 2
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 3 | 2
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 56 | 70
CEREBROVASCULAR DISORDER (Nervous system disorders) | 1 | 2
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 2 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 2 | 2
CEREBRAL ARTERIOSCLEROSIS (Nervous system disorders) | 3 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 22 | 25
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 | 1
CEREBROVASCULAR INSUFFICIENCY (Nervous system disorders) | 1 | 0
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 3 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 2 | 0
HAEMORRHAGIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 3 | 2
NAUSEA (Gastrointestinal disorders) | 4 | 10
APHAGIA (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 3 | 2
COLITIS (Gastrointestinal disorders) | 3 | 5
MELAENA (Gastrointestinal disorders) | 4 | 3
SUBILEUS (Gastrointestinal disorders) | 1 | 1
VOLVULUS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 7 | 8
DIARRHOEA (Gastrointestinal disorders) | 8 | 6
DYSPEPSIA (Gastrointestinal disorders) | 3 | 0
ENTERITIS (Gastrointestinal disorders) | 3 | 0
FAECALOMA (Gastrointestinal disorders) | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 7 | 6
DUODENITIS (Gastrointestinal disorders) | 1 | 0
PERITONITIS (Gastrointestinal disorders) | 2 | 0
SIGMOIDITIS (Gastrointestinal disorders) | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
ANAL FISTULA (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 4
DIVERTICULUM (Gastrointestinal disorders) | 2 | 2
HAEMATEMESIS (Gastrointestinal disorders) | 4 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 2 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 1
PANCREATITIS (Gastrointestinal disorders) | 2 | 6
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 2
RECTAL POLYP (Gastrointestinal disorders) | 1 | 0
ACUTE ABDOMEN (Gastrointestinal disorders) | 2 | 0
COLONIC POLYP (Gastrointestinal disorders) | 2 | 3
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 5 | 4
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 2
ABDOMINAL MASS (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 | 17
DUODENAL ULCER (Gastrointestinal disorders) | 4 | 5
FEMORAL HERNIA (Gastrointestinal disorders) | 1 | 0
GASTRIC POLYPS (Gastrointestinal disorders) | 1 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 7 | 9
INTESTINAL MASS (Gastrointestinal disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 3
DUODENAL FISTULA (Gastrointestinal disorders) | 1 | 0
INTESTINAL POLYP (Gastrointestinal disorders) | 2 | 0
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 | 0
SPIGELIAN HERNIA (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 5 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 2 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 5 | 3
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 2
EROSIVE DUODENITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 4 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 7 | 6
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
PANCREATIC NECROSIS (Gastrointestinal disorders) | 2 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 2
MESENTERIC OCCLUSION (Gastrointestinal disorders) | 0 | 1
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 3 | 1
INTESTINAL INFARCTION (Gastrointestinal disorders) | 2 | 0
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 3 | 1
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 4 | 6
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 | 6
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 | 0
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 3 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
PANCREATITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
PAPILLA OF VATER STENOSIS (Gastrointestinal disorders) | 0 | 2
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 1
HIATUS HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
BOWEL MOVEMENT IRREGULARITY (Gastrointestinal disorders) | 0 | 1
FEMORAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 2
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 21 | 15
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 2
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 1
THROMBOSIS MESENTERIC VESSEL (Gastrointestinal disorders) | 1 | 3
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 1 | 1
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 6 | 6
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 1
VERTIGO (Ear and labyrinth disorders) | 9 | 8
DEAFNESS (Ear and labyrinth disorders) | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 1 | 0
PRESBYACUSIS (Ear and labyrinth disorders) | 1 | 0
MOTION SICKNESS (Ear and labyrinth disorders) | 2 | 0
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 2
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 | 0
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 0 | 1
SEPSIS (Infections and infestations) | 9 | 15
ABSCESS (Infections and infestations) | 1 | 1
CYSTITIS (Infections and infestations) | 1 | 3
FURUNCLE (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 3 | 2
MASTITIS (Infections and infestations) | 0 | 1
RHINITIS (Infections and infestations) | 1 | 0
CARBUNCLE (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 2 | 0
PAROTITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 87 | 83
PYOTHORAX (Infections and infestations) | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 9 | 7
BRONCHITIS (Infections and infestations) | 31 | 30
CELLULITIS (Infections and infestations) | 11 | 22
ERYSIPELAS (Infections and infestations) | 8 | 9
LARYNGITIS (Infections and infestations) | 0 | 2
PARONYCHIA (Infections and infestations) | 2 | 0
URETHRITIS (Infections and infestations) | 0 | 1
ABSCESS JAW (Infections and infestations) | 1 | 0
BACTERAEMIA (Infections and infestations) | 2 | 1
PHARYNGITIS (Infections and infestations) | 1 | 1
TONSILLITIS (Infections and infestations) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 3
APPENDICITIS (Infections and infestations) | 0 | 4
ENDOCARDITIS (Infections and infestations) | 0 | 4
OTITIS MEDIA (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 7 | 6
TUBERCULOSIS (Infections and infestations) | 0 | 3
BRONCHIOLITIS (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 4 | 3
SALMONELLOSIS (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 4 | 8
LUNG INFECTION (Infections and infestations) | 9 | 13
OTITIS EXTERNA (Infections and infestations) | 0 | 2
PYELONEPHRITIS (Infections and infestations) | 3 | 1
SINOBRONCHITIS (Infections and infestations) | 1 | 0
SUPERINFECTION (Infections and infestations) | 0 | 1
ACUTE SINUSITIS (Infections and infestations) | 1 | 0
ECHINOCOCCIASIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 13 | 8
LOBAR PNEUMONIA (Infections and infestations) | 4 | 2
PNEUMONIA VIRAL (Infections and infestations) | 0 | 1
TOOTH INFECTION (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 2 | 0
WOUND INFECTION (Infections and infestations) | 2 | 2
BRONCHITIS VIRAL (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 10 | 6
PERIANAL ABSCESS (Infections and infestations) | 0 | 1
DIABETIC GANGRENE (Infections and infestations) | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 2 | 1
CELLULITIS ORBITAL (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 1
ABSCESS SOFT TISSUE (Infections and infestations) | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 2 | 0
FUNGAL OESOPHAGITIS (Infections and infestations) | 0 | 1
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 3 | 5
HERPES ZOSTER OTICUS (Infections and infestations) | 0 | 1
NOSOCOMIAL INFECTION (Infections and infestations) | 0 | 1
PERITONEAL INFECTION (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 1
SKIN GRAFT INFECTION (Infections and infestations) | 1 | 0
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 | 0
HAEMOPHILUS INFECTION (Infections and infestations) | 1 | 0
PERITONSILLAR ABSCESS (Infections and infestations) | 0 | 1
PSEUDOMONAS INFECTION (Infections and infestations) | 1 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 1
SPINAL CORD INFECTION (Infections and infestations) | 0 | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 | 0
ENDOCARDITIS BACTERIAL (Infections and infestations) | 0 | 1
INFECTED VARICOSE VEIN (Infections and infestations) | 1 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 2
PYELONEPHRITIS CHRONIC (Infections and infestations) | 0 | 3
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 | 1
RETROPERITONEAL ABSCESS (Infections and infestations) | 1 | 0
STREPTOCOCCAL INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 24 | 32
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 3 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 1
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 12
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 4
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 1
AZOTAEMIA (Renal and urinary disorders) | 2 | 1
NEPHRITIS (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 7 | 9
RENAL CYST (Renal and urinary disorders) | 2 | 1
RENAL MASS (Renal and urinary disorders) | 0 | 1
NEPHROPATHY (Renal and urinary disorders) | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 2
BLADDER MASS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 32 | 30
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 2
RENAL ANEURYSM (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 5
NEPHROSCLEROSIS (Renal and urinary disorders) | 2 | 0
BLADDER PROLAPSE (Renal and urinary disorders) | 1 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 6 | 5
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 3
NEPHROPATHY TOXIC (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 3 | 5
NEPHROTIC SYNDROME (Renal and urinary disorders) | 2 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 21 | 10
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 2 | 0
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 | 2
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 4 | 4
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 3 | 2
URINARY BLADDER POLYP (Renal and urinary disorders) | 1 | 0
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 | 0
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0
RENAL ARTERY THROMBOSIS (Renal and urinary disorders) | 1 | 0
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 0 | 1
HOSPITALISATION (Surgical and medical procedures) | 1 | 1
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 | 0
ARTERIOVENOUS SHUNT OPERATION (Surgical and medical procedures) | 1 | 0
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 2 | 5
OBESITY (Metabolism and nutrition disorders) | 0 | 2
ANOREXIA (Metabolism and nutrition disorders) | 3 | 0
CACHEXIA (Metabolism and nutrition disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 21 | 18
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 10
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1
DIABETIC FOOT (Metabolism and nutrition disorders) | 6 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 11 | 8
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 16 | 8
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 3
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 2
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 11 | 19
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 2
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
HYPEROSMOLAR STATE (Metabolism and nutrition disorders) | 0 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
METABOLIC DISORDER (Metabolism and nutrition disorders) | 2 | 0
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 3 | 5
ANAEMIA (Blood and lymphatic system disorders) | 31 | 27
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 1
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2 | 1
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 0 | 1
ANAEMIA VITAMIN B12 DEFICIENCY (Blood and lymphatic system disorders) | 1 | 0
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4 | 5
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 1
PARAPSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 3
DIABETIC ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 | 1
HYPOAESTHESIA FACIAL (Skin and subcutaneous tissue disorders) | 1 | 0
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 0 | 1
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 | 0
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 1
COLPOCELE (Reproductive system and breast disorders) | 0 | 1
CYSTOCELE (Reproductive system and breast disorders) | 0 | 1
RECTOCELE (Reproductive system and breast disorders) | 0 | 2
PROSTATISM (Reproductive system and breast disorders) | 1 | 0
BREAST MASS (Reproductive system and breast disorders) | 2 | 0
PROSTATITIS (Reproductive system and breast disorders) | 1 | 1
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 3
OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 2
CERVIX DISORDER (Reproductive system and breast disorders) | 0 | 1
GENITAL PROLAPSE (Reproductive system and breast disorders) | 1 | 0
UTERINE DISORDER (Reproductive system and breast disorders) | 0 | 1
UTERINE PROLAPSE (Reproductive system and breast disorders) | 2 | 1
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 | 1
PROSTATIC DISORDER (Reproductive system and breast disorders) | 0 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 | 1
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 | 1
UTERINE CERVIX STENOSIS (Reproductive system and breast disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 5 | 4
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 22 | 23
WOUND (Injury, poisoning and procedural complications) | 1 | 1
INJURY (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 3 | 1
CONTUSION (Injury, poisoning and procedural complications) | 3 | 3
CONCUSSION (Injury, poisoning and procedural complications) | 5 | 2
EYE INJURY (Injury, poisoning and procedural complications) | 1 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 1
EXCORIATION (Injury, poisoning and procedural complications) | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 8 | 2
HEAT STROKE (Injury, poisoning and procedural complications) | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 12 | 9
JOINT INJURY (Injury, poisoning and procedural complications) | 2 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 | 5
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 1
DRUG TOXICITY (Injury, poisoning and procedural complications) | 1 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ANIMAL SCRATCH (Injury, poisoning and procedural complications) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 | 5
DEVICE FAILURE (Injury, poisoning and procedural complications) | 1 | 2
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 10 | 7
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 | 0
ILIUM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
RETINAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUTURE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 | 2
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
EYEBALL RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 3 | 3
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 4 | 1
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 2 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 3 | 2
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 1
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 1 | 0
DEVICE DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 3 | 2
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 4 | 1
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 4 | 2
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
HAEMATURIA TRAUMATIC (Injury, poisoning and procedural complications) | 0 | 1
POSTOPERATIVE HERNIA (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 0
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 | 1
CARDIAC VALVE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
CHEMICAL BURN OF SKIN (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 3
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
EXPOSURE TO TOXIC AGENT (Injury, poisoning and procedural complications) | 0 | 1
TRACHEOSTOMY MALFUNCTION (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
DEVICE ELECTRICAL FINDING (Injury, poisoning and procedural complications) | 0 | 3
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 1 | 0
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 2 | 2
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
CARDIAC PACEMAKER MALFUNCTION (Injury, poisoning and procedural complications) | 11 | 3
ARTERIOVENOUS GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 0 | 2
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2
BURSITIS (Musculoskeletal and connective tissue disorders) | 3 | 1
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 | 11
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 4
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 3 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 | 7
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 1
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
GOUTY TOPHUS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 3 | 1
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
METATARSALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 3
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 37 | 24
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 5 | 2
FLOATING PATELLA (Musculoskeletal and connective tissue disorders) | 1 | 0
ACQUIRED CLAW TOE (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 6
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 | 0
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
LOWER LIMB DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 2
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 2 | 2
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 4
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 3
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 3 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 | 4
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 65 | 72
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 4
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 5 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 1
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 4 | 3
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 4 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8 | 5
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 15 | 25
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 4 | 2
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NOCTURNAL DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 20 | 27
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 | 2
PLEURAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 9 | 15
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HILUM MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY AMYLOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 9 | 12
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 5
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
CHEYNE-STOKES RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 21 | 23
PAIN (General disorders) | 0 | 1
DEATH (General disorders) | 5 | 9
POLYP (General disorders) | 0 | 1
CHILLS (General disorders) | 0 | 2
HERNIA (General disorders) | 1 | 2
NODULE (General disorders) | 1 | 0
OEDEMA (General disorders) | 2 | 1
FATIGUE (General disorders) | 4 | 3
MALAISE (General disorders) | 8 | 5
PYREXIA (General disorders) | 6 | 8
ASTHENIA (General disorders) | 8 | 7
EFFUSION (General disorders) | 0 | 1
NECROSIS (General disorders) | 0 | 5
DYSPLASIA (General disorders) | 1 | 0
ENANTHEMA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 75 | 81
SUDDEN DEATH (General disorders) | 70 | 76
ADVERSE EVENT (General disorders) | 0 | 1
CARDIAC DEATH (General disorders) | 1 | 0
ACCIDENTAL DEATH (General disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 4 | 5
GAIT DISTURBANCE (General disorders) | 0 | 1
IMPAIRED HEALING (General disorders) | 1 | 1
LOCALISED OEDEMA (General disorders) | 0 | 1
PERFORATED ULCER (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 8 | 11
ULCER HAEMORRHAGE (General disorders) | 0 | 1
GENERALISED OEDEMA (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 5 | 2
PERIPHERAL COLDNESS (General disorders) | 1 | 0
SUDDEN CARDIAC DEATH (General disorders) | 6 | 11
ADVERSE DRUG REACTION (General disorders) | 1 | 0
IMPLANT SITE HAEMATOMA (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 6 | 5
TEMPERATURE INTOLERANCE (General disorders) | 1 | 0
CATHETER RELATED COMPLICATION (General disorders) | 0 | 1
DRUG CHEMICAL INCOMPATIBILITY (General disorders) | 0 | 1
MECHANICAL COMPLICATION OF IMPLANT (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 8 | 7
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5
LIP NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 10
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
NEOPLASM SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
TONSIL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 7
RECTAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRACHEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
URETHRAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
CARCINOID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
PLEURAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
ABDOMINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12
COLON CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO PLEURA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
RECTAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CERVIX CARCINOMA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RETROPERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MUSCLE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN MEDIASTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MYELOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MALIGNANT FIBROUS HISTIOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
MALIGNANT URINARY TRACT NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
WALDENSTROM'S MACROGLOBULINAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LENTIGO MALIGNA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHRONIC LYMPHOCYTIC LEUKAEMIA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC MYELOID LEUKAEMIA TRANSFORMATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IRBESARTAN (N=2064) | PLACEBO (N=2062)
CARDIAC FAILURE (Cardiac disorders) | 133 | 134
ATRIAL FIBRILLATION (Cardiac disorders) | 108 | 110
HYPOTENSION (Vascular disorders) | 203 | 93
HYPERTENSION (Vascular disorders) | 202 | 252
HEADACHE (Nervous system disorders) | 126 | 138
DIZZINESS (Nervous system disorders) | 262 | 253
DIARRHOEA (Gastrointestinal disorders) | 127 | 89
INFLUENZA (Infections and infestations) | 124 | 111
BRONCHITIS (Infections and infestations) | 176 | 205
NASOPHARYNGITIS (Infections and infestations) | 180 | 174
BACK PAIN (Musculoskeletal and connective tissue disorders) | 132 | 117
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 108 | 104
COUGH (Respiratory, thoracic and mediastinal disorders) | 99 | 117
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 177 | 217
FATIGUE (General disorders) | 108 | 96
CHEST PAIN (General disorders) | 150 | 136
OEDEMA PERIPHERAL (General disorders) | 204 | 205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.